CLINICAL TRIAL: NCT05754385
Title: Effectiveness of Ambulatory Liver Fat Monitoring in Improvement of Hepatic Steatosis in Patients With Non-alcoholic Fatty Liver Disease: a Multi-center Randomized Controlled Trial
Brief Title: Ambulatory Liver Fat Monitoring in Patients With Non-alcoholic Fatty Liver Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Gense Technologies Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKU_EIT_am_liver
Record Dates: First submitted 2023-02-19; First posted 2023-03-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: ambulatory monitoring
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulatory liver fat monitoring (Active Comparator): A novel portable, home-based device called the Gense-EIT liver scan will be given to each participant to practice ambulatory liver fat monitoring
  Interventions: Behavioral: Ambulatory monitoring of liver fat
- Standard of care (Placebo Comparator): Subjects will have follow-up every 6 months by hepatologists for routine care
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Ambulatory monitoring of liver fat — Participants will be given a novel portable, home-based device called the Gense-EIT liver scan the participants and will practice ambulatory liver fat monitoring for 6 months.
  Arms: Ambulatory liver fat monitoring
Behavioral: Standard of care — Subjects will have follow-up every 6 months by hepatologists for routine care
  Arms: Standard of care

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) affects 25% of the global population and causes serious complications, including cirrhosis, hepatocellular carcinoma or mortality. Unfortunately, there are not yet any approved drugs to treatment NAFLD. The only effective means to improve NAFLD is by weight reduction via lifestyle modifications, i.e., diet and physical activity. Most NAFLD patients lack the motivation to initiate and maintain lifestyle modifications. The investigators hypothesize that ambulatory monitoring of liver fat can help NAFLD patients lose more liver fat by motivating them to gain a sense of control over their condition.

DETAILED DESCRIPTION:
As NAFLD is a chronic medical illness, NAFLD patients are not able to receive timely feedback from their effort, and they are often frustrated. Also, living with NAFLD may not cause major perturbations to their usual life, as NAFLD is mostly asymptomatic and patients can easily forget the significance of this condition in the long run. The investigators plan to design a randomized, controlled, non-blinded, multi-centre study to compare the effects of ambulatory liver fat monitoring and standard of care in reduction of liver fat in NAFLD patients. Fibroscan and MRI-PDFF will be used for quantification of hepatic steatosis. Apart from the effect on liver fat, the investigators will also investigate whether ambulatory liver fat monitoring promotes more weight loss and improvement in liver biochemistry.

ELIGIBILITY:
Inclusion Criteria:

* patients with known NAFLD (diagnosed by ultrasonography or other forms of imaging; transient elastography with controlled attenuation parameter >248 dB/m; or liver biopsy) who are managed in the Liver Clinics of Queen Mary Hospital or Tung Wah Hospital
* aged 18-65 years
* without major cognitive impairment - since these subjects would be given simple instructions on using the ambulatory device to measure liver fat at home by themselves

Exclusion Criteria:

* on SGLT-2 inhibitors, GLP-1 agonists, or thiazolidinediones due to their prominent effects on body weight changes
* patients with cirrhosis (defined by imaging features of nodular liver and evidence of portal hypertension, liver stiffness >13 kPa, endoscopically proven gastroesophageal varices, or histological features), with or without ascites
* patients who are pregnant
* patients on special diet or with special dietary requirement (e.g., vegan, gluten free) heavy alcohol use (≥20 grams/ day for women or ≥30 grams/ day for men)
* history of HCC, hepatic resection, or LT
* patients with damaged skin on the abdomen, as this will affect the assessment by the ambulatory liver fat device
* patients with implanted electronic devices
* patients with spinal diseases/ discomfort
* patients with metallic implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with significant hepatic fat change | 6 months
  Efficacy of ambulatory liver fat monitoring versus SOC in achieving significant MRI-PDFF change in NAFLD patients

SECONDARY OUTCOMES:
Percentage of hepatic fat change | 12 months
  Efficacy of ambulatory liver fat monitoring versus SOC in achieving significant MRI-PDFF change in NAFLD patients
Percentage of hepatic fat change | 6 months
  Efficacy of ambulatory liver fat monitoring versus SOC in achieving significant CAP change in NAFLD patients
Percentage of weight change | 6 months
  Efficacy of ambulatory liver fat monitoring versus SOC in achieving significant weight change in NAFLD patients
Percentage of subjects with normalisation of alanine aminotransferase | 6 months
  Efficacy of ambulatory liver fat monitoring versus SOC in achieving normalisation of alanine aminotransferase among NAFLD subjects

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Yi Mak, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Select A State Or Province, China